CLINICAL TRIAL: NCT03559478
Title: Sharp Dissection Versus Monopolar Electrocautery in Primary Total Knee Arthroplasty Performed Under Tourniquet: a Randomized Double Blind Controlled Trial
Brief Title: Sharp Dissection Versus Monopolar Electrocautery in Primary Total Knee Arthroplasty Performed Under Tourniquet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Chloe Scott, Consultant Trauma and Orthopaedic Surgeon, Royal Infirmary of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 244896
Record Dates: First submitted 2018-04-10; First posted 2018-06-18 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Osteo Arthritis Knee; Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Electrocoagulation

STUDY DESIGN:
Intervention Model Description: A total of 70 participants will be randomized in a 1:1 ratio to either Treatment Group 1 (sharp dissection with scalpel plus electrocautery to obvious vessels) or Treatment Group 2 (electrocautery for all dissection) using the sealed opaque envelope randomization technique.
Who Masked: Participant
Masking Description: Patients will be blinded to the intervention as they will be under anaesthetic whilst the procedure is being carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Active Comparator): Sharp dissection with scalpel plus electrocautery to vessels
  Interventions: Procedure: Sharp dissection with scalpel plus electrocautery to vessels
- Treatment Group 2 (Active Comparator): Electrocautery for all dissection
  Interventions: Procedure: Electrocautery for all dissection

INTERVENTIONS:
Procedure: Sharp dissection with scalpel plus electrocautery to vessels — A scalpel will be used for dissection for TKA implantation. Bleeding vessels will be managed as encountered with electrocautery. Electrocautery will not be used for dissection.
  Arms: Treatment Group 1
Procedure: Electrocautery for all dissection — Skin incision will be made with a scalpel, but all other dissection will be performed with electrocautery.
  Arms: Treatment Group 2

SUMMARY:
This study compares the use of sharp dissection with diathermy for the approach to a total knee replacement. Half of the patients will be randomly assigned each intervention.

DETAILED DESCRIPTION:
The approach to the knee to carry out a total knee replacement (TKR) can either be carried out using a scalpel, sharp dissection, or using an electric current to divide tissue, monopoly electrocautery. Reducing blood loss is important. Blood loss can result in anaemia, which has a number of effects including shortness of breath, chest pain and lethargy. Blood loss into a newly replaced knee can also result in pain and stiffness in the joint. Total knee replacements are routinely carried out with a tourniquet inflated, which reduces the blood flow into to leg during the operation. Diathermy is applied to areas of bleeding to stop them from doing so during operations. With the tourniquet inflated, some areas that would bleed when this was deflated may not be noticed and continue to bleed. Using diathermy for the approach would be expected to reduce this bleeding compared to using a scalpel.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee osteoarthritis requiring TKA (total knee arthroplasty)
* Planned for cruciate retaining prosthesis without patella resurfacing
* Patient is able to give informed consent
* Patient resides locally and will be available for follow up

Exclusion Criteria:

* Cardiac pacemaker
* Inflammatory arthropathy
* Tourniquet contraindicated
* Thrombophilia/haemoglobinopathy
* Spinal anaesthetic not possible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
24hr Calculated blood loss | 1 day
  Will be done using the Nadler and Gross formulae

SECONDARY OUTCOMES:
Haemoglobin drop | 1 day
  Haemoglobin drop from day 1 full blood count test
Transfusion requirement | 2 days
  If the patient requires blood transfusion or not
VAS (Visual Analogue Scale) pain score 24 and 48 hrs | 2 days
  Patient's pain score at 24 and 48 hours post-operatively
Range of motion 48hrs and 6 weeks | 6 weeks
  Knee range of motion in degrees at 48 hours and 6 weeks post-operatively
Length of hospital stay | 2 weeks
  Length of inpatient stay in hospital
Improvement in Oxford knee score at 12 months | 12 months
  Oxford Knee Score, designed to assess function and pain after total knee replacement. Scored from 0 (severe knee symptoms with functional limitation) to 60 (absence of pain and limitations)
Adverse events | 12 months
  Any complications encountered

CONTACTS AND LOCATIONS:
Overall Officials: Chloe EH Scott, MD MSc, Principal Investigator — Consultant Trauma and Orthopaedic Surgeon
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No